CLINICAL TRIAL: NCT02135861
Title: An Evaluation of DCE-MRI Measures of Pulmonary Oedema and Vascular Permeability in Healthy Subjects and in Patients With Cardiac Failure: A Methods Validation Study for Evaluation of Novel Treatments Limiting Pulmonary Oedema in Cardiac Failure
Brief Title: A Method Validation Study for Evaluation of Novel Treatments Limiting Pulmonary Oedema in Cardiac Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201137
Record Dates: First submitted 2014-04-24; First posted 2014-05-12 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure, Congestive
Keywords: Acute decompensated heart failure; heart failure; MRI; trpV4 channel inhibitors; pulmonary oedema
MeSH Terms: conditions — Heart Failure; Pulmonary Edema | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): All subjects will undergo MRI scanning conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
  Interventions: Procedure: DCE-MRI scans; Other: Gadobutrol
- Heart failure patients (Experimental): All subjects will undergo DCE-MRI scanning conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 T system.
  Interventions: Procedure: DCE-MRI scans; Other: Gadobutrol
- Acute decompensated heart failure (Experimental): All subjects will undergo DCE-MRI scanning conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 T system
  Interventions: Procedure: DCE-MRI scans; Other: Gadobutrol

INTERVENTIONS:
Procedure: DCE-MRI scans — Subjects will be placed supine in the scanner and will be prepared for intravenous contrast agent administration. The contrast agent is administered using a power injector before imaging.
Other: Gadobutrol — Gadobutrol at a dose less than or equal to 0.1 millimoles per kilogram (mmol/kg) will be given intravenously as a bolus using a power injector.

SUMMARY:
Transient receptor potential vanilloid 4 (TRPV4) channel blockade may be promising in the treatment of pulmonary oedema and dyspnoea in heart failure (HF) and acute decompensated heart failure (ADHF) patients by re-establishing the alveolar septal barrier. Dynamic contrast enhanced (DCE) Magnetic Resonance Imaging (MRI) is an established technique for assessing changes in vascular permeability and interstitial water volume. The aim of this study is to establish the potential utility of DCE-MRI as a novel endpoint for dose ranging and proof of mechanism studies of TRPV4 blockers. The DCE-MRI markers of vascular permeability and pulmonary oedema will be measured in subjects with HF (group 2) and healthy volunteers (HV) (group 1) at rest to determine if there is a difference between the two populations. Apart from this, exercise induced changes relative to rest in interstitial volume and exchange rate will be evaluated in both HV and subjects with HF. Additionally, the capability of DCE-MRI to detect changes in interstitial lung fluid in patients with acute decompensated heart failure (ADHF) (group 3) will be investigated. DCE-MRI markers of pulmonary oedema will be assessed when patients are initially hospitalized with ADHF and subsequently after receiving standard of care treatment to determine whether differences can be detected by this methodology.This study will enrol a sufficient number of subjects to have at least 24 subjects in Group 1 and 2 (group 1:12 HV and group 2: 12 subjects with HF) and atleast 5 subjects in Group 3. For each subject, the MRI data must be of sufficient quality to enable DCE-MRI modelling from 2 Sessions. For group 1 and 2, the subjects will have screening visit and 3 MRI sessions. For the first scanning session, subjects will undergo the baseline procedure. The second imaging session will occur approximately one week later to measure within subject variability. A third imaging session (which will be conducted in 2 visits) will incorporate a bicycle exercise challenge prior to the MRI scan, and this third scan will be performed approximately one to three days after the second imaging session. For group 3: Screening will occur during hospitalization for eligibility. Session 1of MRI will be conducted while the subject is still hospitalized. Session 2 will be conducted within 4 weeks of the first scan, when the signs of pulmonary oedema are considered to be resolved. If a subject's pulmonary oedema has not resolved at Session 2, then the subject will be not be scanned by MRI at Session 2 and will be brought back for Session 3 up to 4 weeks after Session 2 for their second MRI.

ELIGIBILITY:
Inclusion Criteria:

* Male or females over 18 years of age at the time of signing the informed consent.
* Body weight >=50 kilogram (kg) and Body Mass Index (BMI) within the range 18.0-40.0 kilogram/square meter (kg/m^2) (inclusive).
* Able to understand and comply with protocol requirements, instructions and protocol stated restrictions and is willing to take part in the imaging sessions.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Inclusion Criteria for Heart Failure Group (group 2) - Established diagnosis of mild to moderate heart failure of any aetiology with symptoms defined as corresponding to the New York Heart Association (NYHA) class II or III.

Inclusion Criteria for Healthy Volunteer Group (group 1)

- Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, brief physical examination, clinical laboratory tests, and Electrocardiogram (ECG).

Inclusion Criteria for Subjects with ADHF (Group 3)

* Male subjects OR female subjects of non reproductive potential as defined as pre-menopausal females with a documented tubal ligation or hysterectomy, or post-menopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units (MIU)/millilitre (mL) and oestradiol < 40picogram (pg)/mL (< 140 pmol/L) is confirmatory.
* 50 years of age or over at the time of signing the informed consent
* Hospitalized for the management of acute decompensated HF
* Presence of dyspnoea at rest or with minimal activity
* Presence of at least one of the following signs: Tachypnea with respiratory rate >=20 breaths/min or Rales or crackles audible on auscultation
* Chest x-ray with evidence of pulmonary congestion/oedema performed approximately within the last 48 hours (if not available - an additional research CXR may be requested)
* Have received at least one treatment with an intravenous diuretic prior to the first MRI scan
* Body weight >= 50kg and BMI within the range 18-40 kg/m^2 (inclusive)
* Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is willing to take part in the imaging sessions
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion criteria:

Exclusion Criteria for Heart Failure Group

* History of known primary pulmonary disease requiring current medication or other therapy.
* Orthopnoea of sufficient severity to preclude supine scanning as determined at screening.
* Unstable angina within the past 3 months.
* Uncontrolled hypertension (resting systolic Blood Pressure (BP) >160 millimeters of mercury (mmHg) or resting diastolic BP >100 mmHg).
* Resting hypoxia while breathing room air (Saturation of Oxygen [SaO2] <88%). Exclusion Criteria for Healthy Volunteer Group and Heart Failure Groups
* Current smoker, defined as having smoked in the preceding 6 months.
* Contraindication for MRI scanning (as assessed by local MRI safety questionnaire) which includes but not limited to: Intracranial aneurysm clips or other metallic objects; Intra-orbital metal fragments that have not been removed ; Pacemakers or other implanted cardiac rhythm management devices and non-MRI compatible heart valves; Inner ear implants; and History of claustrophobia.
* Pregnant females as determined by positive urine human chorionic gonadotropin (HCG) test at screening or any scanning session.
* Positive test for drugs of abuse, not due to current prescription drugs as determined by the GSK Medical Monitor and principal investigator (PI), and alcohol screen.
* Estimated Creatinine Clearance (Cockcroft-Gault) <60 millilitre (mL)/minute.

Exclusion Criteria for Subjects with ADHF (Group 3)

* End-stage heart failure defined as requiring left ventricular assist devices, intra-aortic balloon pump or any type of mechanical support
* Chronic or intermittent renal support therapy (hemodialysis, ultrafiltration, or peritoneal dialysis)
* Ongoing or planned intravenous diuretic treatment within 1 hour of MRI scan appointment
* History of known primary pulmonary disease requiring current medication or other therapy
* Orthopnoea of sufficient severity to preclude supine scanning (as determined by a 15-minute test of lying supine with or without the use of oxygen)
* Contraindication for MRI scanning (as assessed by local MRI safety questionnaire), which includes but is not limited to: Intracranial aneurysm clips (except Sugita) or other metallic objects OR intra-orbital metal fragments that have not been removed OR pacemakers or other implanted cardiac rhythm management devices and non-MRI compatible heart valves OR inner ear implants OR history of claustrophobia
* Estimated creatinine clearance (Cockcroft-Gault) <40mL/minute
* Contraindication to MRI contrast agents
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden(a significant radiation burden being defined as 10 millisieverts (mSv) in addition to natural background radiation, in the previous 3 years including the dose from this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included healthy volunteers (HV, group 1), participants (par) with heart failure (HF, group 2) and participants with acute decompensated heart failure (ADHF, group 3) who were hospitalized with evidence of pulmonary edema and received standard of care treatment.
Pre-assignment Details: Dynamic Contrast Enhanced-Magnetic Resonance Imaging (DCE-MRI) markers were used to measure vascular permeability and pulmonary edema in HV and par. with HF. Forty one par. were enrolled and 36 entered the study. Three par. did not continue due to habitus and 2 par. did not participate as they required clinical investigations.
Groups:
- Healthy Volunteers: Healthy volunteers were placed in supine position under the scanner and intravenous contrast agent was administered. Contrast agent was administered as a bolus using a power injector during the dynamic series. MRI scanning was conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
- Heart Failure Participants: Heart failure participants were placed in supine position under the scanner and intravenous contrast agent was administered. Contrast agent was administered as a bolus using a power injector during the dynamic series. MRI scanning was conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
- Acute Decompensated Heart Failure Participants: Acute Decompensated Heart Failure participants following hospitalization due to pulmonary oedema was placed in supine position under the scanner and intravenous contrast agent was administered. Contrast agent was administered as a bolus using a power injector during the dynamic series. MRI scanning was conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
Period: Overall Study
Arm/Group | Healthy Volunteers | Heart Failure Participants | Acute Decompensated Heart Failure Participants
Started | 21 | 12 | 3
Completed | 21 | 12 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Heart Failure Participants | Acute Decompensated Heart Failure Participants | Total
Number analyzed (Participants) | 21 | 12 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (18.66) | 67.8 (13.42) | 79.3 (4.93) | 66.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 19 | 10 | 2 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 0 | 1 | 0 | 1
  White | 21 | 11 | 3 | 35

OUTCOME MEASURES:

1. Primary Outcome: Interstitial Volume (ve) in Heart Failure Participants and Healthy Volunteers at Baseline
Description: Interstitial volume (ve) was measured by DCE-MRI. ve for total lung, left lung, right lung, left lung apical, left lung basal, right lung apical, right lung basal has been presented. Session 1 values were considered as Baseline values.
Time Frame: Day 1
Population: The Evaluable Population will include participants in safety population who are 40 years and older .The safety Population includes all enrolled participants who have initiated Session 1 DCE-MRI scan
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Healthy Volunteers | Heart Failure Participants
Number analyzed (Participants) | 17 | 12
Liter
  Total lung | 0.4946 (0.0362) | 0.3346 (0.0325)
  Left lung | 0.5078 (0.0349) | 0.3253 (0.0317)
  Right lung | 0.4960 (0.0417) | 0.3395 (0.0371)
  Left lung apical | 0.4952 (0.0339) | 0.3188 (0.0306)
  Left lung basal | 0.5349 (0.0397) | 0.3350 (0.0362)
  Right lung apical | 0.4865 (0.0392) | 0.3506 (0.0352)
  Right lung basal | 0.5045 (0.0444) | 0.3297 (0.0390)
Statistical Analysis 1: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0029, ANOVA — estimates of total lung; Mean Difference (Final Values) = 0.1600, 95% CI 2-sided [0.0600 to 0.2600]; Ve was fitted using a repeat measure ANOVA model with terms including participant population (HF or HV), visit (i.e. sessions), interaction of participant population and visit, with participant ID as block of the repeat factor
Statistical Analysis 2: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0007, ANOVA — estimates of left lung; Mean Difference (Final Values) = 0.1825, 95% CI 2-sided [0.0855 to 0.2795]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0093, ANOVA — estimates of right lung; Mean Difference (Final Values) = 0.1565, 95% CI 2-sided [0.0419 to 0.2711]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0007, ANOVA — estimates of left lung apical; Mean Difference (Final Values) = 0.1764, 95% CI 2-sided [0.0823 to 0.2704]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0010, ANOVA — estimates of left lung basal; Mean Difference (Final Values) = 0.1999, 95% CI 2-sided [0.0894 to 0.3103]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0159, ANOVA — estimates of right lung apical; Mean Difference (Final Values) = 0.1360, 95% CI 2-sided [0.0276 to 0.2443]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Healthy Volunteers vs Heart Failure Participants; Test type: Other; p = 0.0064, ANOVA — estimates of right lung basal; Mean Difference (Final Values) = 0.1748, 95% CI 2-sided [0.0535 to 0.2961]; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Exchange Rate (Ktrans) in Heart Failure Participants and Healthy Volunteers at Baseline
Description: Exchange rate (Ktrans) was measured by DCE-MRI. Ktrans for total lung, left lung, right lung, left lung apical, left lung basal, right lung apical, right lung basal has been presented. Session 1 values were considered as Baseline values.
Time Frame: Day 1
Population: The Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Heart Failure Participants | Healthy Volunteers
Number analyzed (Participants) | 12 | 17
Liter/minute
  Total lung | 0.2216 (0.0298) | 0.2353 (0.0273)
  Left lung | 0.2309 (0.0256) | 0.2173 (0.0236)
  Right lung | 0.2216 (0.0338) | 0.2474 (0.0309)
  Left lung apical | 0.2166 (0.0265) | 0.2161 (0.0244)
  Left lung basal | 0.2621 (0.0270) | 0.2225 (0.0249)
  Right lung apical | 0.2166 (0.0355) | 0.2528 (0.0326)
  Right lung basal | 0.2313 (0.0329) | 0.2431 (0.0301)
Statistical Analysis 1: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.7381, ANOVA — estimates of total lung; Mean Difference (Final Values) = -0.0137, 95% CI 2-sided [-0.0968 to 0.0695]; Ktrans was fitted using a repeat measure ANOVA model with terms including participant population (HF or HV), visit (i.e. sessions), interaction of participant population and visit, with participant ID as block of the repeat factor
Statistical Analysis 2: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.6992, ANOVA — estimates of left lung; Mean Difference (Final Values) = 0.0136, 95% CI 2-sided [-0.0580 to 0.0852]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.5778, ANOVA — estimates of right lung; Mean Difference (Final Values) = -0.0258, 95% CI 2-sided [-0.1201 to 0.0684]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.9899, ANOVA — estimates of left lung apical; Mean Difference (Final Values) = 0.0005, 95% CI 2-sided [-0.0738 to 0.0747]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.2912, ANOVA — estimates of left lung basal; Mean Difference (Final Values) = 0.0396, 95% CI 2-sided [-0.0360 to 0.1153]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.4592, ANOVA — estimates of right lung apical; Mean Difference (Final Values) = -0.0362, 95% CI 2-sided [-0.1355 to 0.0631]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.7936, ANOVA — estimates of right lung basal; Mean Difference (Final Values) = -0.0118, 95% CI 2-sided [-0.1036 to 0.0800]; [other analysis details as in outcome 2, analysis 1]

3. Primary Outcome: Interstitial Volume (ve) in Heart Failure Participants and Healthy Volunteers Before and Following Exercise
Description: Interstitial volume (ve) was measured by DCE-MRI. ve for total lung, left lung, right lung, left lung apical, left lung basal, right lung apical, right lung basal before and following exercise has been presented.
Time Frame: Day 11
Population: The Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Heart Failure Participants | Healthy Volunteers
Number analyzed (Participants) | 12 | 17
Liter
  Pre-exercise; Total lung | 0.4353 (0.0335) | 0.3205 (0.0292)
  Post-exercise; Total lung | 0.4568 (0.0307) | 0.3140 (0.0263)
  Pre-exercise; Left lung | 0.4487 (0.0311) | 0.3121 (0.0267)
  Post-exercise; Left lung | 0.4832 (0.0266) | 0.3055 (0.0228)
  Pre-exercise; Right lung | 0.4361 (0.0357) | 0.3294 (0.0311)
  Post-exercise; Right lung | 0.4534 (0.0355) | 0.3274 (0.0298)
  Pre-exercise; Left lung apical | 0.4272 (0.0335) | 0.3126 (0.0289)
  Post-exercise; Left lung apical | 0.4449 (0.0257) | 0.2986 (0.0216)
  Pre-exercise; Left lung basal | 0.4890 (0.0318) | 0.3114 (0.0272)
  Post-exercise; Left lung basal | 0.5310 (0.0323) | 0.3173 (0.0276)
  Pre-exercise; Right lung apical | 0.4343 (0.0378) | 0.3387 (0.0324)
  Post-exercise; Right lung apical | 0.4504 (0.0358) | 0.3393 (0.0301)
  Pre-exercise; Right lung basal | 0.4400 (0.0347) | 0.3206 (0.0301)
  Post-exercise; Right lung basal | 0.4591 (0.0367) | 0.3133 (0.0308)
Statistical Analysis 1: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0156, ANOVA — estimates of total lung- Pre-exercise; Mean Difference (Final Values) = 0.1148, 95% CI 2-sided [0.0236 to 0.2061]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0026, ANOVA — estimates of left lung- Pre-exercise; estimates of left lung- Pre-exercise; Mean Difference (Final Values) = 0.1366, 95% CI 2-sided [0.0523 to 0.2209]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0328, ANOVA — estimates of right lung- Pre-exercise; Mean Difference (Final Values) = 0.1067, 95% CI 2-sided [0.0094 to 0.2040]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0158, ANOVA — estimates of left lung apical-Pre-exercise; Mean Difference (Final Values) = 0.1145, 95% CI 2-sided [0.0235 to 0.2056]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0002, ANOVA — estimates of left lung basal-Pre-exercise; Mean Difference (Final Values) = 0.1776, 95% CI 2-sided [0.0917 to 0.2635]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0658, ANOVA — estimates of right lung apical-Pre-exercise; Mean Difference (Final Values) = 0.0956, 95% CI 2-sided [-0.0067 to 0.1979]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0150, ANOVA — estimates of right lung basal-Pre-exercise; Mean Difference (Final Values) = 0.1194, 95% CI 2-sided [0.0251 to 0.2137]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0015, ANOVA — estimates of total lung-Post-exercise; Mean Difference (Final Values) = 0.1428, 95% CI 2-sided [0.0598 to 0.2259]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p < .0001, ANOVA — estimates of left lung-Post-exercise; Mean Difference (Final Values) = 0.1776, 95% CI 2-sided [0.1057 to 0.2496]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0114, ANOVA — estimates of right lung-Post-exercise; Mean Difference (Final Values) = 0.1260, 95% CI 2-sided [0.0308 to 0.2212]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0002, ANOVA — estimates of left lung apical-Post-exercise; Mean Difference (Final Values) = 0.1464, 95% CI 2-sided [0.0774 to 0.2153]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p < .0001, ANOVA — estimates of left lung basal-Post-exercise; Mean Difference (Final Values) = 0.2137, 95% CI 2-sided [0.1266 to 0.3008]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0250, ANOVA — estimates of right lung apical-Post-exercise; Mean Difference (Final Values) = 0.1111, 95% CI 2-sided [0.0151 to 0.2071]; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.0052, ANOVA — estimates of right lung basal-Post-exercise; Mean Difference (Final Values) = 0.1458, 95% CI [0.0475 to 0.2442]; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Exchange Rate (Ktrans) in Heart Failure Participants and Healthy Volunteers Before and Following Exercise
Description: Exchange rate (Ktrans) was measured by DCE-MRI. Ktrans for total lung, left lung, right lung, left lung apical, left lung basal, right lung apical, right lung basal before and following exercise has been presented.
Time Frame: Day 11
Population: The Evaluable Population
Measure: Least Squares Mean (Standard Error); unit: Liter/minute
Arm/Group | Heart Failure Participants | Healthy Volunteers
Number analyzed (Participants) | 12 | 17
Liter/minute
  Pre-exercise; Total lung | 0.2044 (0.0281) | 0.2567 (0.0247)
  Post-exercise; Total lung | 0.1841 (0.0221) | 0.2108 (0.0190)
  Pre-exercise; Left lung | 0.2102 (0.0285) | 0.2525 (0.0245)
  Post-exercise; Left lung | 0.1785 (0.0200) | 0.1986 (0.0172)
  Pre-exercise; Right lung | 0.2034 (0.0299) | 0.2550 (0.0263)
  Post-exercise; Right lung | 0.1926 (0.0269) | 0.2114 (0.0226)
  Pre-exercise; Left lung apical | 0.1856 (0.0293) | 0.2459 (0.0253)
  Post-exercise; Left lung apical | 0.1621 (0.0199) | 0.1780 (0.0167)
  Pre-exercise; Left lung basal | 0.2552 (0.0296) | 0.2630 (0.0254)
  Post-exercise; Left lung basal | 0.2060 (0.0227) | 0.2185 (0.0196)
  Pre-exercise; Right lung apical | 0.1934 (0.0281) | 0.2440 (0.0243)
  Post-exercise; Right lung apical | 0.1892 (0.0267) | 0.2141 (0.0224)
  Pre-exercise; Right lung basal | 0.2181 (0.0319) | 0.2593 (0.0281)
  Post-exercise; Right lung basal | 0.2052 (0.0284) | 0.2081 (0.0238)
Statistical Analysis 1: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.1730, ANOVA — estimates of total lung-Pre-exercise; Mean Difference (Final Values) = -0.0524, 95% CI 2-sided [-0.1292 to 0.0244]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.2704, ANOVA — estimates of left lung-Pre-exercise; Mean Difference (Final Values) = -0.0423, 95% CI 2-sided [-0.1196 to 0.0349]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.2072, ANOVA — estimates of right lung-Pre-exercise; Mean Difference (Final Values) = -0.0515, 95% CI 2-sided [-0.1334 to 0.0303]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.1307, ANOVA — estimates of left lung apical-Pre-exercise; Mean Difference (Final Values) = -0.0603, 95% CI 2-sided [-0.1398 to 0.0191]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.8427, ANOVA — estimates of left lung basal-Pre-exercise; Mean Difference (Final Values) = -0.0078, 95% CI 2-sided [-0.0879 to 0.0722]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.1848, ANOVA — estimates of right lung apical-Pre-exercise; Mean Difference (Final Values) = -0.0506, 95% CI 2-sided [-0.1269 to 0.0257]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.3408, ANOVA — estimates of right lung basal-Pre-exercise; Mean Difference (Final Values) = -0.0413, 95% CI 2-sided [-0.1286 to 0.0461]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.3682, ANOVA — estimates of total lung-Post-excercise; Mean Difference (Final Values) = -0.0267, 95% CI 2-sided [-0.0866 to 0.0332]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.4531, ANOVA — estimates of left lung-Post-excercise; Mean Difference (Net) = -0.0201, 95% CI 2-sided [-0.0744 to 0.0342]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.5970, ANOVA — estimates of right lung-Post-excercise; Mean Difference (Final Values) = -0.0188, 95% CI 2-sided [-0.0909 to 0.0533]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.5472, ANOVA — estimates of left lung apical-Post-excercise; Mean Difference (Final Values) = -0.0159, 95% CI 2-sided [-0.0693 to 0.0375]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.6793, ANOVA — estimates of left lung basal-Post-excercise; Mean Difference (Final Values) = -0.0125, 95% CI 2-sided [-0.0742 to 0.0491]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.4806, ANOVA — estimates of right lung apical-Post-excercise; Mean Difference (Final Values) = -0.0249, 95% CI 2-sided [-0.0964 to 0.0466]; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Heart Failure Participants vs Healthy Volunteers; Test type: Other; p = 0.9379, ANOVA — estimates of right lung basal-Post-excercise; Mean Difference (Final Values) = -0.0029, 95% CI 2-sided [-0.0789 to 0.0731]; [other analysis details as in outcome 2, analysis 1]

5. Primary Outcome: Change in Interstitial Volume (ve) in ADHF Participants
Description: Interstitial volume (ve) was measured by DCE-MRI. Three participants underwent 3 DCE-MRI scans. The data has been presented for individual participant in each session. The data presented below is only for total lung.
Time Frame: Up to Week 8
Population: The safety population will include all enrolled participants who have initiated at least one session of DCE-MRI or Lung Ultrasound Scan
Measure: Number; unit: Liter
Arm/Group | Acute Decompensated Heart Failure Participants
Number analyzed (Participants) | 3
Liter
  Par.1; Session 1 | 0.794
  Par.1; Session 2 | 0.9577
  Par. 2; Session 1 | 0.5086
  Par. 2; Session 2 | 0.4018
  Par. 3; Session 1 | 0.354
  Par. 3; Session 2 | 0.6356
  Par. 3 Session 3 | 0.6083

6. Primary Outcome: Change in Exchange Rate (Ktrans) in ADHF Participants
Description: Exchange rate (Ktrans) was measured by DCE-MRI. Three participants underwent 3 DCE-MRI scans. The data has been presented for individual participant in each session. The data presented below is only for total lung.
Time Frame: Up to Week 8
Population: The Safety Population
Measure: Number; unit: Liter/minute
Arm/Group | Acute Decompensated Heart Failure Participants
Number analyzed (Participants) | 3
Liter/minute
  Par.1; Session 1 | 0.4524
  Par.1; Session 2 | 0.5306
  Par. 2; Session 1 | 0.3018
  Par. 2; Session 2 | 0.1952
  Par. 3; Session 1 | 0.1602
  Par. 3; Session 2 | 0.4304
  Par. 3 Session 3 | 0.4264

7. Secondary Outcome: Assessment of Intra-subject Variability in Ve Between Session 1 and Session 2 of DCE-MRI
Description: Coefficient of variation (percentage) of intra-subject variability in Ve between Session 1 and Session 2 for total lung has been presented.
Time Frame: Day 1 (Session 1) and Day 9 (Session 2)
Population: The Evaluable Population
Measure: Number; unit: Percentage
Arm/Group | Heart Failure Participants | Healthy Volunteers
Number analyzed (Participants) | 12 | 17
Percentage | 20.5 | 14.1

8. Secondary Outcome: Assessment of Intra-subject Variability in Ktrans Between Session 1 and Session 2 of DCE-MRI
Description: Coefficient of variation (percentage) of intra-subject variability in Ktrans between Session 1 and Session 2 for total lung has been presented.
Time Frame: Day 1 (Session 1) and Day 9 (Session 2)
Population: The Evaluable Population
Measure: Number; unit: Percentage
Arm/Group | Heart Failure Participants | Healthy Volunteers
Number analyzed (Participants) | 12 | 17
Percentage | 32.4 | 41.3

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and AEs related to study procedure were planned to be collected from the start of study procedure and up to last visit (Up to Week 8)
Description: SAEs and non-serious AEs related to study procedure were planned to be reported for Safety Population
Groups:
- Heart Failure Patients: Heart failure participants were placed in supine position under the scanner and intravenous contrast agent was administered. Contrast agent was administered as a bolus using a power injector during the dynamic series. MRI scanning was conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
- Acute Decompensated Heart Failure: Acute Decompensated Heart Failure participants following hospitalization due to pulmonary oedema was placed in supine position under the scanner and intravenous contrast agent was administered. Contrast agent was administered as a bolus using a power injector during the dynamic series. MRI scanning was conducted by experienced radiographers and radiologists in the nominated scanning sites, using a 1.5 Tesla (T) system.
Arm/Group | Healthy Volunteers | Heart Failure Patients | Acute Decompensated Heart Failure
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 0/17 | 0/12 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02135861/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT02135861/SAP_001.pdf